CLINICAL TRIAL: NCT02819856
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of SPI-1005 in Cystic Fibrosis (CF) Patients With Acute Pulmonary Exacerbation (APE) Receiving IV Tobramycin at Risk for Ototoxicity
Brief Title: SPI-1005 for Prevention and Treatment of Tobramycin Induced Ototoxicity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sound Pharmaceuticals, Incorporated (Industry)
Collaborators: Medical University of South Carolina (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-3005-501
Record Dates: First submitted 2016-06-16; First posted 2016-06-30 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Ototoxicity
Keywords: Ebselen; Tinnitus; Hearing Loss; Vertigo; Cystic Fibrosis; Pulmonary Exacerbation; Tobramycin; Safety; Pharmacokinetics; Pharmacodynamics; Aminoglycoside; SPI-1005; Efficacy; Pharmacogenomics; Ototoxicity
MeSH Terms: conditions — Ototoxicity; Tinnitus; Hearing Loss; Vertigo; Cystic Fibrosis | interventions — ebselen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SPI-1000 Capsule 0mg Ebselen Placebo (Placebo Comparator): 0mg Ebselen SPI-1000 bid po x 21d
  Interventions: Drug: Placebo
- SPI-1005 Ebselen 200mg Capsule x1 (Experimental): 200mg SPI-1005 bid po x 21d Low Dose Arm
  Interventions: Drug: SPI-1005 Ebselen 200mg Capsule x1
- SPI-1005 Ebselen 200mg Capsule x2 (Experimental): 400mg SPI-1005 bid po x 21d Mid Dose Arm
  Interventions: Drug: SPI-1005 Ebselen 200mg Capsule x2
- SPI-1005 Ebselen 200mg Capsule x3 (Experimental): 600mg SPI-1005 bid po x 21d High Dose Arm
  Interventions: Drug: SPI-1005 Ebselen 200mg Capsule x3

INTERVENTIONS:
Drug: Placebo — 0 mg SPI-1005 bid po x 21d
  Other Names: SPI-1000
  Arms: SPI-1000 Capsule 0mg Ebselen Placebo
Drug: SPI-1005 Ebselen 200mg Capsule x1 — 200 mg SPI-1005 bid po x21d
  Other Names: SPI-1005 Low Dose
  Arms: SPI-1005 Ebselen 200mg Capsule x1
Drug: SPI-1005 Ebselen 200mg Capsule x2 — 400 mg SPI-1005 bid po x 21d
  Other Names: SPI-1005 Mid Dose
  Arms: SPI-1005 Ebselen 200mg Capsule x2
Drug: SPI-1005 Ebselen 200mg Capsule x3 — 600 mg SPI-1005 bid po x 21d
  Other Names: SPI-1005 High Dose
  Arms: SPI-1005 Ebselen 200mg Capsule x3

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of SPI-1005 treatment in CF patients with active pulmonary exacerbation that are receiving an IV course of tobramycin, determined by comparing hearing assessments, spirometry, Pharmacokinetic (PK), Physical Exam, Adverse Events (AEs) and Labs baseline to post-treatment.

The secondary objectives of this study are to determine Pharmacogenomics and Pharmacodynamics of SPI-1005.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled study to evaluate the safety, and efficacy of SPI-1005 in Cystic Fibrosis patients with Acute Pulmonary Exacerbation receiving intravenous tobramycin at risk for ototoxicity. All patients will undergo baseline testing and have their severity of lung function, sensorineural hearing loss, tinnitus and vertigo determined before the start of SPI-1005 treatment. SPI-1005 treatment will start within first two days of IV tobramycin treatment and be administered concomitantly. At the end of the 21-day course of SPI-1005 and 28 days following the cessation of SPI-1005, patients will have their hearing loss, tinnitus and vertigo reassessed. Assessments may also include additional audiometric and pulmonary testing, and additional follow-up testing.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis patients about to receive IV tobramycin for acute pulmonary exacerbation.
* Voluntarily consent to participate in the study.
* Females of childbearing potential should be using and committed to continue using one of the following acceptable birth control methods:
* Sexual abstinence (inactivity) for 14 days prior to screening through study completion; or IUD in place for at least 3 months prior to study through study completion; or Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening through study completion; or Stable hormonal contraceptive for at least 3 months prior to study through study completion.
* Ability to perform all behavioral tests as indicated.

Exclusion Criteria:

* Current use or within 60 days prior to study enrollment the following IV ototoxic medications: aminoglycoside antibiotics (gentamicin, tobramycin, amikacin, streptomycin); platinum-containing chemotherapies (cisplatin, carboplatin, oxaliplatin); or loop diuretic (furosemide).
* History of idiopathic sensorineural hearing loss, otosclerosis, or vestibular schwannoma.
* History of middle ear or inner ear surgery.
* Current conductive hearing loss or middle ear effusion.
* Significant cardiovascular, hepatic, renal, hematologic, endocrine, immunologic, or psychiatric disease.
* History of hypersensitivity or idiosyncratic reaction to compounds related to ebselen.
* Participation in another investigational drug or device study within 30 days prior to study enrollment.
* Female patients who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with sensorineural hearing loss as a measure of safety and efficacy of SPI-1005 | 7 weeks
  Determination of sensorineural hearing loss using pure-tone audiometry
Distortion Product Otoacoustic Emissions | 7 weeks
  Changes in hearing thresholds using pure-tone audiometry with extended high frequency testing
Speech discrimination | 7 weeks
  Change in Words in noise test (WINT) score
Tinnitus severity | 7 weeks
  Changes in Tinnitus Functional Index (TFI) score
Vertigo severity | 7 weeks
  vertigo symptom scale
Changes in lung function | 7 weeks
  Evaluation of lung function using FEV1
Trough Level of SPI-1005 at 200, 400, and 600 mg Ebselen po bid x 21d | 7 weeks
  Plasma ebselen and major metabolite quantified in plasma by LC-MS/MS

SECONDARY OUTCOMES:
Pharmacogenomics | 5 weeks
  Pharmacogenomics analysis will explore SPI-1005 as an inducer of gene expression for Nrf2, glutathione peroxidase-1, hemeoxygenase-1, and thioredoxin class of redox proteins.
Pharmacodynamics of Nrf2 | 5 weeks
  Explore SPI-1005 on the level of Nrf2 by PCR
Pharmacodynamics of Glutathione, cysteine and cystine | 5 weeks
  Explore SPI-1005 on the level of Glutathione, cysteine and cystine measured in µM.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kil, MD, Study Chair — SOUND PHARMACEUTICALS, INC.
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Takumida M, Popa R, Anniko M. Free radicals in the guinea pig inner ear following gentamicin exposure. ORL J Otorhinolaryngol Relat Spec. 1999 Mar-Apr;61(2):63-70. doi: 10.1159/000027643. PMID 10095194
- [Background] Kil J, Pierce C, Tran H, Gu R, Lynch ED. Ebselen treatment reduces noise induced hearing loss via the mimicry and induction of glutathione peroxidase. Hear Res. 2007 Apr;226(1-2):44-51. doi: 10.1016/j.heares.2006.08.006. Epub 2006 Oct 6. PMID 17030476
- [Background] Flume PA, Mogayzel PJ Jr, Robinson KA, Goss CH, Rosenblatt RL, Kuhn RJ, Marshall BC; Clinical Practice Guidelines for Pulmonary Therapies Committee. Cystic fibrosis pulmonary guidelines: treatment of pulmonary exacerbations. Am J Respir Crit Care Med. 2009 Nov 1;180(9):802-8. doi: 10.1164/rccm.200812-1845PP. Epub 2009 Sep 3. PMID 19729669
- [Background] Gu R, Longenecker RJ, Homan J, Kil J. Ebselen attenuates tobramycin-induced ototoxicity in mice. J Cyst Fibros. 2021 Mar;20(2):271-277. doi: 10.1016/j.jcf.2020.02.014. Epub 2020 Mar 5. PMID 32147183
- [Background] Harruff EE, Kil J, Ortiz MGT, Dorgan D, Jain R, Poth EA, Fifer RC, Kim YJM, Shoup AG, Flume PA. Ototoxicity in cystic fibrosis patients receiving intravenous tobramycin for acute pulmonary exacerbation: Ototoxicity following tobramycin treatment. J Cyst Fibros. 2021 Mar;20(2):288-294. doi: 10.1016/j.jcf.2020.11.020. Epub 2020 Dec 16. PMID 33341407